CLINICAL TRIAL: NCT07227298
Title: AN INTERVENTIONAL OPEN-LABEL PHASE 1B/2 STUDY TO EVALUATE THE SAFETY, PHARMACOKINETICS, AND PRELIMINARY EFFICACY OF PF-08634404 IN COMBINATION WITH DIFFERENT ANTICANCER AGENTS IN PARTICIPANTS WITH ADVANCED SOLID TUMORS
Brief Title: A Study to Learn About the Study Medicine Called PF-08634404 in Combination With Different Anticancer Agents in Advanced Cancers
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: C6461020; 2025-523526-40-00 (EU CTIS Number)
Record Dates: First submitted 2025-11-07; First posted 2025-11-12 (Actual); Last update posted 2025-11-12 (Actual); Status verified 2025-11

CONDITIONS: Advanced/Metastatic Non-Small Cell Lung Cancer; Carcinoma, Non-Small Cell Lung; Non-Small Cell Lung Cancer
Keywords: non-small cell lung cancer; NSCLC; advanced solid tumors; metastatic non-small cell lung cancer; locally advanced non-small cell lung cancer; squamous non-small cell lung cancer; non-squamous non-small cell lung cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- PF-08634404 + Sigvotatug Vedotin (Part A) (Experimental): Participants will receive PF-08634404 in combination with Sigvotatug Vedotin.
  Interventions: Biological: PF-08634404; Biological: Sigvotatug Vedotin
- PF-08634404 + Combination Agent 1 (Part B) (Experimental): Participants will receive PF-08634404 in combination with other anticancer agent as per protocol.
  Interventions: Biological: PF-08634404; Biological: Combination Agent 1

INTERVENTIONS:
Biological: PF-08634404 — -Concentrate for solution for infusion
  Other Names: SSGJ-707
Biological: Sigvotatug Vedotin — -Powder for concentrate for solution for infusion. Single use vial
  Other Names: SGN-B6A; PF-08046047
  Arms: PF-08634404 + Sigvotatug Vedotin (Part A)
Biological: Combination Agent 1 — -Powder for concentrate for solution for infusion. Single use vial.
  Arms: PF-08634404 + Combination Agent 1 (Part B)

SUMMARY:
This study is being done to learn more about a new medicine called PF-08634404 and how it works when used with other cancer medicines in people who have advanced solid tumors. An advanced solid tumor is a type of cancer that has spread beyond its original location and cannot be removed by surgery or cured with standard treatments.

To join in the study, participants must:

* Be 18 years or older
* Participants with advanced non-small cell lung cancer (NSCLC), a type of lung cancer that has spread

The study will look at:

* Whether PF-08634404 is safe to use with other cancer medicines.
* What side effects may happen. A side effect is anything the medicine does to your body that is not part of treating your disease.
* Whether the combination of PF-08634404 and other cancer medicines can help treat solid tumors.

The study has different parts, each testing PF-08634404 with a different cancer medicine:

* Part A will test PF-08634404 with a medicine called sigvotatug vedotin.
* Part B of the study will look at how well the new medicine PF-08634404 works when used together with another medicine.

Participants will receive the study medicines through an intravenous (IV) infusion (injected into the vein) at the study clinic. All treatments will take place at clinical trial sites, where trained medical staff will monitor participants during and after each visit.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically confirmed locally advanced (Stage IIIB/IIIC) or metastatic (Stage IV) squamous or non-squamous NSCLC and are not a candidate for complete surgical resection and curative concurrent/sequential chemoradiotherapy
* PD-L1 status available
* Part B only: PD-L1 ≥ TPS 1%
* Measurable disease based on RECIST v1.1 per investigator.
* Eastern Cooperative Oncology Group performance status of 0 or 1.
* Adequate organ function

Exclusion Criteria:

* Participants with known AGAs including EGFR, ALK and ROS1, NTRK, BRAF, and MET
* History of another malignancy within 3 years before the first dose of study intervention, or any evidence of residual disease from a previously diagnosed malignancy
* Known active CNS lesions, including brainstem, meningeal, or spinal cord metastases or compression
* Leptomeningeal disease
* Active autoimmune diseases requiring systemic treatment within the past 2 years
* Previous systemic anti-tumor therapy for locally advanced, unresectable, or metastatic NSCLC
* Previous treatment with immunotherapy (exception is (neo)adjuvant anti-PD-(L)1), ADCs containing MMAE payload, systemic anti-angiogenic therapy, or prior radiotherapy to the lung within 6 months of first dose of study intervention

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 162 (Estimated)
Dates: Start 2025-11-17 (Estimated); Primary Completion 2029-03-08 (Estimated); Study Completion 2033-08-23 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Treatment Emergent Adverse Events (AEs) and Serious Adverse Events (SAEs) | Through 90 days after the last study intervention; Up to approximately 5 years
  AEs as characterized by type, frequency, severity (as graded by NCI CTCAE version 5.0), timing, seriousness, and relationship to study intervention.
Phase I: Number of participants with dose limiting toxicity (DLT) | Through 90 days after the last study intervention; Up to approximately 5 years
  Dose limiting toxicity based on dose limiting toxicity evaluable participants. The number of participants who experienced DLTs during the DLT observation period.
Phase 2: Confirmed Objective Response Rate (ORR) per RECIST v1.1 by investigator | Up to approximately 5 Years
  ORR is defined as the proportion of participants with a Best Overall Response (BOR) of confirmed Complete Response (CR) or confirmed Partial Response (PR) per RECIST v1.1.

SECONDARY OUTCOMES:
Phase I: Confirmed ORR per RECIST v1.1 by investigator | Up to approximately 5 Years
  ORR is defined as the proportion of participants with a Best Overall Response (BOR) of confirmed Complete Response (CR) or confirmed Partial Response (PR) per RECIST v1.1.
Disease Control Rate (DCR) per RECIST v1.1 by investigator | Up to approximately 5 years
  DCR by investigator assessment is defined as the proportion of participants with CR or PR with confirmation, or Stable Disease (SD) by investigator assessment per RECIST version 1.1.
Duration of Response (DOR) per RECIST v1.1 by investigator | Up to approximately 5 years
  DOR is defined as the time from the first documentation of objective response (CR or PR that is subsequently confirmed) to the date of first documented disease progression per RECIST v1.1 or death due to any cause, whichever occurs first.
Progression Free Survival (PFS) per RECIST v1.1 by investigator | Up to approximately 5 years
  Progression-free survival is defined as the time from the date of randomization to the date of the first documentation of objective PD assessed by investigator per RECIST v1.1, or death due to any cause, whichever occurs first.
Number of Participants With Clinical Laboratory Abnormalities | Through 90 days after the last study intervention; Up to approximately 5 years
Pharmacokinetics (PK): Serum concentration of PF-08634404 with anticancer agents | Up to 37 days after the last dose of treatment
  To characterize the pharmacokinetics (PK) of PF-08634404 with anticancer agents.
Incidence of Anti-Drug Antibody (ADA) against PF-08634404 with anticancer agents | Up to 37 days after the last dose of treatment
  To characterize the immunogenicity of PF-08634404 with anticancer agents.

OTHER OUTCOMES:
Overall Survival (OS) | Up to approximately 5 years
  Overall survival defined as the time from the date of randomization to the date of death due to any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.